CLINICAL TRIAL: NCT04191772
Title: The Impact of Structured Exercise on Physical Fitness, Sedentary Time, Brain Volume, Cognitive, Health-related and Immunological Parameters in Multiple Sclerosis.
Brief Title: The Impact of Training on Sitting Time and Brain Volumes in Multiple Sclerosis.
Acronym: EXIMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Bert Op't Eijnde, Principal Investigator, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXIMS
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Multiple Sclerosis
Keywords: Sedentary time; Exercise; Brain volume; Health-related variables; Immunological variables; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will receive an intervention (exercise program) or no intervention (sedentary control group). Participants will be persons with MS and healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- MS - training goal 1 (Experimental): Persons with Multiple Sclerosis (PwMS) with a 'poor VO2max', a 'fair VO2max' with no running experience and a 'good VO2max' with no running experience (VO2max values according to V.H. Heyward, Advanced Fitness Assessment and Exercise Prescription, Fifth Edition, 2006, Champaign, IL: Human Kinetics) will receive an exercise intervention existing of home-based running sessions. Participants of the first training group will be trained to run continuously for 45 minutes.
  Interventions: Other: Periodized, home-based running program
- HC - training goal 1 (Experimental): Healthy control (HC) persons with a 'poor VO2max', a 'fair VO2max' with no running experience and a 'good VO2max' with no running experience (VO2max values according to V.H. Heyward, Advanced Fitness Assessment and Exercise Prescription, Fifth Edition, 2006, Champaign, IL: Human Kinetics) will receive an exercise intervention existing of home-based running sessions. Participants of the first training group will be trained to run continuously for 45 minutes.
  Interventions: Other: Periodized, home-based running program
- MS - training goal 2 (Experimental): PwMS with a 'fair VO2max' and running experience, a 'good VO2max and running experience', an 'excellent VO2max' and a 'superior VO2max' (VO2max values according to V.H. Heyward, Advanced Fitness Assessment and Exercise Prescription, Fifth Edition, 2006, Champaign, IL: Human Kinetics) will receive an exercise intervention existing of home-based running sessions. Participants of the second training group will be trained to run continuously for 75 minutes.
  Interventions: Other: Periodized, home-based running program
- HC - training goal 2 (Experimental): HC with a 'fair VO2max' and running experience, a 'good VO2max and running experience', an 'excellent VO2max' and a 'superior VO2max' (VO2max values according to V.H. Heyward, Advanced Fitness Assessment and Exercise Prescription, Fifth Edition, 2006, Champaign, IL: Human Kinetics) will receive an exercise intervention existing of home-based running sessions. Participants of the second training group will be trained to run continuously for 75 minutes.
  Interventions: Other: Periodized, home-based running program
- MS - sedentary control group (No Intervention): Twenty PwMS will receive no intervention, only usual care.
- HC - sedentary control group (No Intervention): Twenty HC will receive no intervention, only usual care.

INTERVENTIONS:
Other: Periodized, home-based running program — All participants will perform a home-based supervised exercise training program. Participants will receive weekly training instructions using a smartphone-based heart rate monitor application (Polar® app). Training sessions will involve running and the design of the training program will be based on linear periodization, where aerobic capacity is built firstly through a period of high-volume/low-intensity training before the proportion of high-intensity training is increased. The total duration of the exercise program will be 12 months with three weekly training sessions. Training progression will be dependent on initial VO2max values and running experience. VO2max classification is based on reference values described in V.H. Heyward, Advanced Fitness Assessment and Exercise Prescription, Fifth Edition, 2006, Champaign, IL: Human Kinetics.
  Arms: HC - training goal 1; HC - training goal 2; MS - training goal 1; MS - training goal 2

SUMMARY:
The current study aims to investigate whether persons with Multiple Sclerosis (PwMS) compensate training time with more sedentary time and consequently blunt training effects. The second aim will be to investigate the effect of a structured training program on specific brain volumes and cognitive variables.

DETAILED DESCRIPTION:
Multiple Sclerosis is a progressive, autoimmune, neurodegenerative disorder of the central nervous system (CNS) that predominantly affects young to middle-aged adults. It is characterized by a chronic inflammatory process that causes demyelination, axonal damage and white matter lesions across the CNS. Furthermore, evidence also indicates grey matter (GM) atrophy which has been reported to be significantly correlated with both clinical and cognitive deterioration. Clinical manifestations include spasticity, tremor, paralysis, walking difficulties and cognitive abnormalities. Due to these primary disease symptoms, persons with MS (PwMS) appear to be susceptible to a sedentary lifestyle and inactivity, which consequently increases the risk of other important, health-related secondary deficits including respiratory, metabolic and cardiac dysfunction. These deficits further contribute to a decrease in cardiorespiratory fitness and quality of life (QoL), thereby causing a vicious circle of decreased exercise tolerance, greater disability and increased inactivity. Since pharmacological treatment has little impact on these secondary deficits, exercise therapy has become an important aspect of the treatment of MS.

Hence, exercise therapy interventions in MS have been studied extensively and have already been proven to significantly improve cardiorespiratory fitness, muscle strength, balance, fatigue, cognition, quality of life, respiratory function and brain volumes. Moreover, a dose-response relationship has been reported for functional variables such as strength and endurance capacity. As such, high intensity interval training (HIIT) probably is exerts superior effects compared to traditional low/moderate intensity continuous training (MICT). However and in contrast with other populations, effects of HIIT on important health-related variables such as body composition, blood pressure and blood lipid profiles are less evident. Possibly, PwMS do not reach the exercise intensities required to improve such factors due to cardiovascular autonomic dysfunction, leading to impaired carotid baroreflex control, attenuated elevations in blood pressure and disturbed increases in heart rate, and abnormal muscle energy metabolism. Moreover, higher intensities might hamper longer-term implementation in real life, as an inverse relation between exercise intensity and training adherence has already been reported.

Training periodization (alternating HIIT and MICT) offers a solution to overcome the barrier of adherence and concurrently augmenting training effects, but in contrast to other populations, the addition of a lower intensity training component does still not improve health-related variables. Therefore, other approaches are warranted. Recently, evidence is growing that sedentary time is an important health risk factor, independent of the (dis)practice of structured exercise. Hence, PwMS possibly compensate training effects with even more sedentary time, in addition to an already sedentary lifestyle as mentioned previously. As such, addressing sedentary time might be an interesting new approach to counteract the health-related deficits in PwMS. Therefore, the present study explores the impact of a structured exercise program on sedentary time and health-related variables.

Furthermore, a secondary aim of the current project is to investigate the effect of a periodized training program on brain volumes and cognitive function. Recent evidence of physical training effects on cognitive variables is contradictory. So for exercise intervention studies that studied the latter only used short-term and laboratory-based training programs and included exercise modalities (type, intensity, duration) that are difficult to compare. Interestingly, a recent short-term randomized controlled trial reported superior effects of HIIT on cognitive functions compared to MICT. Hence, the current study aims to investigate the impact of a long-term, home-based training program with HIIT-components on cognitive variables.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis according to the McDonald criteria (Relaps remitting)
* Written informed consent
* Medical safety screening

Exclusion Criteria:

* Contra-indications to participate in moderate to high intensity exercise
* Contra-indications to undergo magnetic resonance imaging (pacemaker/defibrillator or wires other than sternal wires, insulin pumps, metal foreign bodies, deep brain stimulator, cerebral aneurysm clips, cochlear implant, magnetic dental implant, drug infusion device)
* Medication changes in the last month before the start of the intervention
* Following or plan to follow a weight reduction program
* Pregnancy
* Participation in another study
* Acute MS exacerbation < 3 months prior to the start of the study
* EDSS score > 4
* Consumption of more than 20 alcohol units/week
* No daily internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of steps per day | Before start of the training program
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Number of steps per day | Week 1 of the training program
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Number of steps per day | Week 24 of the training program
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Number of steps per day | Week 48 of the training program
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Number of steps per day | 3 months after the training program
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Sitting time | Before start of the training program
  Sedentary behaviour will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Sitting time | Week 1 of the training program
  Sedentary behaviour will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Sitting time | Week 24 of the training program
  Sedentary behaviour will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Sitting time | Week 48 of the training program
  Sedentary behaviour will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Sitting time | 3 months after the training program
  Sedentary behaviour will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Standing time | Before start of the training program
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Standing time | Week 1 of the training program
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Standing time | Week 24 of the training program
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Standing time | Week 48 of the training program
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Standing time | 3 months after the training program
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Stepping time | Before start of the training program
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Stepping time | Week 1 of the training program
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Stepping time | Week 24 of the training program
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Stepping time | Week 48 of the training program
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).
Stepping time | 3 months after the training program
  Physical activity will be measured with the ActivPAL3TM activity monitor (PAL Technologies Ltd, Glasgow, UK).

SECONDARY OUTCOMES:
Blood pressure | Baseline
  Systolic, diastolic and mean arterial blood pressure will be measured 4 times at 5-min intervals after an initial resting period of 10min, using an electronic sphygmomanometer (Omron®, Omron Healthcare, IL, USA) from the dominant arm and documented as the mean value of the final 3 measurements.
Blood pressure | Week 48 of the training program
  Systolic, diastolic and mean arterial blood pressure will be measured 4 times at 5-min intervals after an initial resting period of 10min, using an electronic sphygmomanometer (Omron®, Omron Healthcare, IL, USA) from the dominant arm and documented as the mean value of the final 3 measurements.
Resting heart rate | Baseline
  Resting heart rate will be measured 4 times at 5-min intervals after an initial resting period of 10min, using an electronic sphygmomanometer (Omron®, Omron Healthcare, IL, USA) from the dominant arm and documented as the mean value of the final 3 measurements.
Resting heart rate | Week 48 of the training program
  Resting heart rate will be measured 4 times at 5-min intervals after an initial resting period of 10min, using an electronic sphygmomanometer (Omron®, Omron Healthcare, IL, USA) from the dominant arm and documented as the mean value of the final 3 measurements.
Total calorie intake | Baseline
  Participants will record all food and beverages consumed over seven consecutive days and from this the total calorie intake is calculated.
Total calorie intake | Week 12 of the training program
  Participants will record all food and beverages consumed over seven consecutive days and from this the total calorie intake is calculated.
Total calorie intake | Week 24 of the training program
  Participants will record all food and beverages consumed over seven consecutive days and from this the total calorie intake is calculated.
Total calorie intake | Week 48 of the training program
  Participants will record all food and beverages consumed over seven consecutive days and from this the total calorie intake is calculated.
Total calorie intake | 3 months after the training program
  Participants will record all food and beverages consumed over seven consecutive days and from this the total calorie intake is calculated.
Macronutrient content | Baseline
  Participants will record all food and beverages consumed over seven consecutive days and from this the macronutrient content is calculated.
Macronutrient content | Week 12 of the training program
  Participants will record all food and beverages consumed over seven consecutive days and from this the macronutrient content is calculated.
Macronutrient content | Week 24 of the training program
  Participants will record all food and beverages consumed over seven consecutive days and from this the macronutrient content is calculated.
Macronutrient content | Week 48 of the training program
  Participants will record all food and beverages consumed over seven consecutive days and from this the macronutrient content is calculated.
Macronutrient content | 3 months after the training program
  Participants will record all food and beverages consumed over seven consecutive days and from this the macronutrient content is calculated.
Participation - Ghent Participation Scale (GPS) | Baseline
  The GPS is a generic instrument including both objective and all relevant subjective variables resulting in one score, already proven to be valid to rate participation in MS.
Participation - Ghent Participation Scale (GPS) | Week 48 of the training program
  The GPS is a generic instrument including both objective and all relevant subjective variables resulting in one score, already proven to be valid to rate participation in MS.
Mobility - MS walking scale (MSWS-12) | Baseline
  The MSWS-12 is a 12-item self-assessment scale which measures the impact of MS on mobility, which showed the ability of a running program to reduce impact of MS on walking ability in a previous pilot RCT by our research group
Mobility - MS walking scale (MSWS-12) | Week 48 of the training program
  The MSWS-12 is a 12-item self-assessment scale which measures the impact of MS on mobility, which showed the ability of a running program to reduce impact of MS on walking ability in a previous pilot RCT by our research group
Fatigue - Modified Fatigue Impact scale (MFIS) | Before start of the intervention
  To evaluate the impact of structured training on fatigue, the Modified Fatigue Impact Scale (MFIS) will be used, which is the recommended questionnaire for research related to fatigue by the Multiple Sclerosis Council for Clinical guidelines. In the MFIS, the perceived impact of fatigue on physical, cognitive and psychosocial functioning of the past 4 weeks is assessed.
Fatigue - Modified Fatigue Impact scale (MFIS) | Week 1 of the intervention
  To evaluate the impact of structured training on fatigue, the Modified Fatigue Impact Scale (MFIS) will be used, which is the recommended questionnaire for research related to fatigue by the Multiple Sclerosis Council for Clinical guidelines. In the MFIS, the perceived impact of fatigue on physical, cognitive and psychosocial functioning of the past 4 weeks is assessed.
Fatigue - Modified Fatigue Impact scale (MFIS) | Week 12 of the training program
  To evaluate the impact of structured training on fatigue, the Modified Fatigue Impact Scale (MFIS) will be used, which is the recommended questionnaire for research related to fatigue by the Multiple Sclerosis Council for Clinical guidelines. In the MFIS, the perceived impact of fatigue on physical, cognitive and psychosocial functioning of the past 4 weeks is assessed.
Fatigue - Modified Fatigue Impact scale (MFIS) | Week 24 of the training program
  To evaluate the impact of structured training on fatigue, the Modified Fatigue Impact Scale (MFIS) will be used, which is the recommended questionnaire for research related to fatigue by the Multiple Sclerosis Council for Clinical guidelines. In the MFIS, the perceived impact of fatigue on physical, cognitive and psychosocial functioning of the past 4 weeks is assessed.
Fatigue - Modified Fatigue Impact scale (MFIS) | Week 48 of the training program
  To evaluate the impact of structured training on fatigue, the Modified Fatigue Impact Scale (MFIS) will be used, which is the recommended questionnaire for research related to fatigue by the Multiple Sclerosis Council for Clinical guidelines. In the MFIS, the perceived impact of fatigue on physical, cognitive and psychosocial functioning of the past 4 weeks is assessed.
Fatigue - Modified Fatigue Impact scale (MFIS) | 3 months after the training program
  To evaluate the impact of structured training on fatigue, the Modified Fatigue Impact Scale (MFIS) will be used, which is the recommended questionnaire for research related to fatigue by the Multiple Sclerosis Council for Clinical guidelines. In the MFIS, the perceived impact of fatigue on physical, cognitive and psychosocial functioning of the past 4 weeks is assessed.
Cognition - Spatial Recall test (SPART) | Baseline
  The SPART is a visuospatial learning and delayed recall test, where a checkerboard with seven checkers in specified places is presented for 10sec to the participants who have to place the checkers back on a blank checkerboard immediately after and after another 30min. The total score is a sum of the correct checkers. This has been shown to be one of the most sensitive measures for detecting memory impairments in PwMS and showed improved performance after a running program in a previous pilot RCT of our research group
Cognition - Spatial Recall test (SPART) | Week 48 of the training program
  The SPART is a visuospatial learning and delayed recall test, where a checkerboard with seven checkers in specified places is presented for 10sec to the participants who have to place the checkers back on a blank checkerboard immediately after and after another 30min. The total score is a sum of the correct checkers. This has been shown to be one of the most sensitive measures for detecting memory impairments in PwMS and showed improved performance after a running program in a previous pilot RCT of our research group
Cognition - Symbol Digit Modalities Test (SDMT) | Baseline
  The SDMT is a test of information processing speed (PS) in which participants need to combine as many symbols with the accompanying numbers as possible in 90 seconds. The SDMT has been found to be a reliable and valid test in MS and a responder definition of approximating 4 points or 10% in magnitude SDMT change was recommended.
Cognition - Symbol Digit Modalities Test (SDMT) | Week 48 of the training program
  The SDMT is a test of information processing speed (PS) in which participants need to combine as many symbols with the accompanying numbers as possible in 90 seconds. The SDMT has been found to be a reliable and valid test in MS and a responder definition of approximating 4 points or 10% in magnitude SDMT change was recommended.
Body weight | Baseline
  Body weight is determined using a digital-balanced weighting scale to the nearest 0.1kg
Body weight | Week 48 of the training program
  Body weight is determined using a digital-balanced weighting scale to the nearest 0.1kg
Height | Baseline
  Body height is measured to the nearest 0.1cm using a wall-mounted Harpenden stadiometer, with participants barefoot
Height | Week 48 of the training program
  Body height is measured to the nearest 0.1cm using a wall-mounted Harpenden stadiometer, with participants barefoot
DEXA (Dual Energy X-Ray) | Baseline
  body fat mass and lean tissue mass using Dual Energy X-ray Absorptiometry
DEXA (Dual Energy X-Ray) | Week 48 of the training program
  body fat mass and lean tissue mass using Dual Energy X-ray Absorptiometry
Coordination - timed tandem walk (TTW) | Baseline
  Participants will have to walk in a straight line with one foot immediately in front of the other (heel to toe), while the arms are kept down at the side. Time to complete 3 meter will be monitored.
Coordination - timed tandem walk (TTW) | Week 48 of the training program
  Participants will have to walk in a straight line with one foot immediately in front of the other (heel to toe), while the arms are kept down at the side. Time to complete 3 meter will be monitored.
Oxygen uptake (VO2) | Baseline
  Cardiopulmonary exercise test on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VO2 is collected breath-by-breath and averaged every ten seconds.
Oxygen uptake (VO2) | Week 48 of the training program
  Cardiopulmonary exercise test on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VO2 is collected breath-by-breath and averaged every ten seconds.
Carbon dioxide output (VCO2) | Baseline
  Cardiopulmonary exercise test on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VCO2 is collected breath-by-breath and averaged every ten seconds.
Carbon dioxide output (VCO2) | Week 48 of the training protocol
  Cardiopulmonary exercise test on on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VCO2 is collected breath-by-breath and averaged every ten seconds.
Minute ventilation (VE) | Baseline
  Cardiopulmonary exercise test on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VE is collected breath-by-breath and averaged every ten seconds.
Minute ventilation (VE) | Week 48 of the training protocol
  Cardiopulmonary exercise test on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VE is collected breath-by-breath and averaged every ten seconds.
Equivalents for oxygen uptake (VE/VO2) | Baseline
  Cardiopulmonary exercise test on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VE/VO2 is collected breath-by-breath and averaged every ten seconds.
Equivalents for oxygen uptake (VE/VO2) | Week 48 of the training protocol
  Cardiopulmonary exercise test on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VE/VO2 is collected breath-by-breath and averaged every ten seconds.
Equivalents for carbon dioxide production (VE/VCO2) | Baseline
  Cardiopulmonary exercise test on on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VE/VCO2 is collected breath-by-breath and averaged every ten seconds.
Equivalents for carbon dioxide production (VE/VCO2) | Week 48 of the training program
  Cardiopulmonary exercise test on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis VE/VCO2 is collected breath-by-breath and averaged every ten seconds.
Tidal volume (Vt) | Baseline
  Cardiopulmonary exercise test on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis Vt is collected breath-by-breath and averaged every ten seconds.
Tidal volume (Vt) | Week 48 of the training program
  Cardiopulmonary exercise test on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis Vt is collected breath-by-breath and averaged every ten seconds.
Breathing frequency (BF) | Baseline
  Cardiopulmonary exercise test on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis BF is collected breath-by-breath and averaged every ten seconds.
Breathing frequency (BF) | Week 48 of the training protocol
  Cardiopulmonary exercise test on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis BF is collected breath-by-breath and averaged every ten seconds.
Respiratory gas exchange ratio (RER) | Baseline
  Cardiopulmonary exercise test on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis RER is collected breath-by-breath and averaged every ten seconds.
Respiratory gas exchange ratio (RER) | Week 48 of the training program
  Cardiopulmonary exercise test on a bicycle ergometer is performed. With the aid of continuous pulmonary gas exchange analysis RER is collected breath-by-breath and averaged every ten seconds.
Cardiorespiratory fitness (CRF) | Baseline
  CRF will be measured with a maximal cardiopulmonary exercise test on a bicycle ergometer.
Cardiorespiratory fitness (CRF) | Week 48 of the training program
  CRF will be measured with a maximal cardiopulmonary exercise test on a bicycle ergometer.
Lipidomic profile | Baseline
  Blood analysis
Lipidomic profile | Week 48 of the training program
  Blood analysis
Brain volumes | Baseline
  MRI scan
Brain volumes | Week 48 of the training program
  MRI scan
PBMC subset parameters | Baseline
  flow cytometry analysis of immune cell subsets in peripheral blood-derived mononuclear cells (PBMCs)
PBMC subset parameters | Week 48 of the training program
  flow cytometry analysis of immune cell subsets in peripheral blood-derived mononuclear cells (PBMCs)
serum cytokines | Baseline
  cytokine levels are measured by ELISA on serum derived from peripheral blood samples
serum cytokines | Week 48 of the training program
  cytokine levels are measured by ELISA on serum derived from peripheral blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Bert Op 't Eijnde, Prof. dr., Study Chair — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium

REFERENCES:
- [Derived] Nieste I, Spaas J, Franssen WMA, Asch PV, Savelberg HHCM, Eijnde BO. The effect of a structured running exercise intervention on non-exercise physical activity and sedentary behaviour in persons with mild Multiple Sclerosis and healthy controls. J Act Sedentary Sleep Behav. 2023 Dec 4;2(1):29. doi: 10.1186/s44167-023-00037-1. PMID 40217416